CLINICAL TRIAL: NCT07142109
Title: Physical Therapist and Patient Perspectives on Emotional Support in Physical Therapy Rehabilitation for Injured Soldiers: An Empirical Investigation of Needs, Facilitators, and Barriers in Providing Body-Mind Support
Brief Title: Exploring Physical Therapists and Wounded Soldiers' Perceptions Toward Integrating Emotional Elements Into Rehabilitation
Status: Recruiting | Type: Observational
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Other Study IDs: UHaifa 334/24
Record Dates: First submitted 2025-07-16; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-07

CONDITIONS: Rehabilitation Programs

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to examine the perceptions, attitudes, and knowledge of physical therapists regarding the integration of emotional support into the rehabilitation of wounded soldiers. It further aims to determine the patients perceptions of their own rehabilitation needs, what motivates them and what acts as barriers to their motivation. Lastly, it aims to explore the physical therapists perceptions as to what enhances or hinders patients motivation for rehabilitation success.

DETAILED DESCRIPTION:
A mixed-methods approach will be used. A survey of Physical therapists working with wounded soldiers (n ≈ 100) will includes personal and professional factors and role perception, empathy, burnout and compassion. Additionally, interviews with Physical therapists and wounded soldiers (n ≈ 28) will explore factors they perceive to influence motivation for physical rehabilitation and successful recovery. All participants will receive an explanation of the research before taking part and will be asked to indicate their consent (for the survey) or sign a consent form (for the interviews). For the quantitative section, descriptive statistics will be used to process and present the data for the research variables. Hypothesis testing will be conducted using parametric or non-parametric goodness-of-fit tests, depending on the distribution of data across research measures. The significance level will be set at p < 0.05. All statistical analyses will be performed using SPSS software, version 22.

For the qualitative section, thematic analysis of the semi-structured interviews will be conducted using Interpretative Phenomenological Analysis.

ELIGIBILITY:
Inclusion Criteria:

* physical therapists who currently work with, or have worked with, injured servicemen in public or private rehabilitation settings.
* Injured servicemen between the ages of 18-35.

Exclusion Criteria:

* Physical therapists with more than one year of professional experience.
* Injured servicemen exclude those who suffered traumatic brain injury

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: Physical therapists will be recruited through advertisements in social media forums, in dedicated physical therapy groups, at relevant conferences in the field, and through non profits that cater to physical therapists. Injured servicemen will also be recruited through online forums, and through snowball sampling. All participants will reside in Israel.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
personal and professional characteristics | Nov 2024 - Dec 2025
  questionnaire we created that includes: gender, age, education, clinical specialty, number of patients seen per week, place of work, participation in training workshops

SECONDARY OUTCOMES:
Role perception questionnaire | Nov 2024 - Dec 2025
  As part of the survey, the Physician Belief Scale will be asked - 14 point questionnaire where participants respond on a likert scale 1 - 5, agree to disagree. Lower scores indicate higher biopsychosocial attitudes.

OTHER OUTCOMES:
Interviews with physical therapists and wounded soldiers | May 2025 - March 2026
  one hour semi structured interviews
Empathy questionnaire | Nov 2024 - Dec 2025
  As part of the survey, the Interpersonal Reactivity Index questionnaire will be asked. The scale comprises 28 questions and 4 subscales (Perspective Taking, Fantasy, Empathic Concern, Personal Distress) and participants respond on a 5- point Likert scale ranging from 1 (does not describe me well) to 5 (describes me very well). The sclae is calculated according to each subscale, and higher scores reflect greater self-reported levels of the corresponding empathy subscale.
Burnout questionnaire | Nov 2024 - Dec 2025
  As part of the survey, the Professional Quality of Life Scale will be used. The scale is 30 questions and 3 subscales (Compassion Satisfaction, Burnout, Secondary Traumatic Stress) and participants respond on a 5-point Likert scale ranging from 1 (never) to 5 (very often). Scores are calculated by summing the scores for each subcategory. Higher scores indicate a higher measure of that specific subcategory.
Compassion Questionnaire | Nov 2024 - Dec 2025
  As part of the survey, compassion levels will be measured using the the Self-Compassion Scale-Short Form. The scale comprises 12 questions and participants respond on a 5-point Likert scale ranging from 0 (almost never) to 4 (almost always). After the necessary questions are reversed, the total mean score is calculated. Higher total score indicates a greater self-compassion

CONTACTS AND LOCATIONS:
Locations (1):
- Haifa University, Haifa, Israel